CLINICAL TRIAL: NCT05592288
Title: The Impact of a Mobile Application Designed for Adults at Risk of Developing Diabetes on Following the Mediterranean Diet Plan, Physical Activity and Metabolic Parameters: a Study Protocol for a Randomized Controlled Trial
Brief Title: The Impact of a Mobile Application Designed for Adults at Risk of Developing Diabetes
Acronym: MobileApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İbrahim TOPUZ, Lecturer (PhD student), Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TDK-2022-6085
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus Risk; PreDiabetes
Keywords: Diabetes Mellitus Risk; PreDiabetes; Mobile application; Physical activity; Mediterranean Diet; Metabolic variables
MeSH Terms: conditions — Prediabetic State; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study protocol was drawn up for a single center, single-blind (participant), pretest-posttest, follow-up, parallel group (1:1 ratio) randomized controlled trial.
Who Masked: Participant
Masking Description: Single-blind (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The study universe will consist of adults of the ages 45-65 who have received a diagnosis of prediabetes and are registered at the Family Health Center No. 9. PREDIABE-TR mobile app usage (six months).
  Interventions: Other: PREDIABE-TR mobile app.
- Control grup (No Intervention): The study universe will consist of adults of the ages 45-65 who have received a diagnosis of prediabetes and are registered at the Family Health Center No. 9. Routine practice (Brochures of the Public Health Directorate, Mobile apps of the Ministry of Health, etc.)

INTERVENTIONS:
Other: PREDIABE-TR mobile app. — * Module 1: Personal data Containing data on the participant's age, gender, telephone number, email and perception of his/her health (bad, so-so, good, very good).
  * Module 2: Medical history of the participant In this module, the participants tick the items that apply to themselves or their first-degree relatives by marking the conditions in their medical history that may increase the risk of prediabetes. Additionally, in line with the recommendations of the Turkish Association of Endocrinology and Metabolism, this module contains the Finnish Diabetes Type-2 Risk Score (FINDRISK) which assesses an individual's risk of diabetes.
  * Module 3: Healthy lifestyle behaviors The sub-sections of the module are devoted to nutrition, height-weight-body mass index (BMI) and physical activity.
  Arms: Intervention group

SUMMARY:
Aim: The aim of this study is to determine whether a prediabetes mobile application (PREDIABE-TR) designed in Turkish to inform and advise individuals at risk of developing diabetes about healthy eating and physical exercise can make a difference in the participants' eating according to the Mediterranean Diet Plan, or in their physical activity and other diabetes-related metabolic parameters.

Methods: A total of 120 adults at risk of developing diabetes will be assigned into an experimental and a control group by means of Stratified Permuted Block Randomization. The adults in the experimental group will be using the PREDIABE-TR mobile application for a period of 6 months. Over the same period, the control group will use the Turkish Nutrition Guide and the Diabetes Checklists mobile application distributed by the Turkish Ministry of Health. At the end of the six-month period, a review will be made of the diabetes metabolic data, physical activity levels and the Mediterranean Diet eating behaviors. At the same time, an assessment will be made of the control group's use of the mobile application with the help of the Mobile Application Usability Scale. Statistical data will be analyzed using the Statistical Package for the Social Sciences program.

Discussion: The benefits of interventions to promote a healthy lifestyle are evident in terms of preventing a transition from prediabetes to diabetes and maintaining present status. The current novel coronavirus pandemic has clearly shown the advantages of and necessity for remote interventions. In this study, we will attempt to determine whether or not the use of the PREDIABE-TR mobile application can promote a healthy lifestyle and achieve a reduced risk of diabetes.

Impact: This study will serve to provide evidence of the practicality, acceptability and cost effectiveness of various applications (such as mobile apps) that can be an alternative to face-to-face consultation and other medical practices. This alternative can be suggested to policy- and decision-makers. Such applications can also be considered preventive strategies.

DETAILED DESCRIPTION:
Hypotheses

Our hypotheses were formulated in line with Population-Intervention-Comparison-Outcome-Study; significance was set at 0.05 (Higgins et al., 2019). In addition to standard applications, the intervention group will be using the PREDIABE-TR mobile app. The control group will only use standard applications. In this context, our research hypotheses are the following:

H1a: When compared with the control group, the eating behaviors with regard to adopting the Mediterranean Diet of prediabetic adults using the PREDIABE-TR app will be at a higher level.

H1b: When compared with the control group, the physical activity (MET, number of steps) of prediabetic adults using the PREDIABE-TR app will be at a higher level.

H1c: When compared with the control group, the metabolic parameters (A1C, Impaired Fasting Glucose, Impaired Glucose Tolerance of prediabetic adults using the PREDIABE-TR app will be at lower levels.

H1d: When compared with the control group, prediabetic adults using the PREDIABE-TR app will lose more weight.

ELIGIBILITY:
Inclusion criteria

* Individuals to be included will be those who: are prediabetic (Impaired Fasting Glucose =100-125 mg/dl-mmol/L, A1C=5.7%-6.4% or Impaired Glucose Tolerance=140-190 mg/dl-mmol/L),
* are active Android/phone operating system cell phone users,
* are not pregnant or have any malignancy,
* have no hearing or vision impairment,
* are at least primary school graduates and fluent in Turkish.

Exclusion criteria

* Individuals who have a diagnosis of diabetes or are using an insulin pump or oral antidiabetic agents,
* have vision impairment,
* are pregnant,
* have any condition that precludes engaging in physical activity,
* have psychiatric issues or problems with communicating, will be excluded.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Mediterranean Diet Adherence Screener-MEDAS) | Change 6 months from baseline
  The Turkish validity and reliability studies for MEDAS.
International Physical Activity Questionnaire (IPAQ) | Change 6 months from baseline
  The IPAQ International Physical Activity Questionnaire-Short Form.
Metabolic Measurements | Change 6 months from baseline
  The participants' A1C, fasting blood glucose values will be measured. The A1C Measurement represents a 3-month mean value The A1C testing does not require fasting conditions. The blood sample can be taken at any time of day. Over the period of the study, the A1C result the participant has obtained from being tested at any health facility will be taken from the personal health system records.
Blood Glucose Measurement | Change 6 months from baseline
  The researcher will measure the participants' blood glucose with a Roche Accu-Chek® perform nano device. A minimum eight-hour fasting period will be taken as a criterion for fasting blood glucose; a postprandial blood glucose test will be administered 2 hours after a meal.

SECONDARY OUTCOMES:
Height-Weight Measurement and Body Mass Index | Change 6 months from baseline
  The researcher will measure the individuals' height and weight with calibrated devices. BMI will be calculated with the formula: weight (kg)/height (m2) (TEMD, Obesity Diagnosis and Treatment Guidelines, 2019).
Mobile App Usability and Usage Assessment Scale | 6th month
  Three measures developed before to assess the usability and usage of a mobile application will be used. The validity and reliability study for the scales was performed for Turkish.
Mobile Application Usability Scale | 6th month
  This is a measure used to assess and understand how the mobile app can be improved and how it may be made more user-friendly. The scale is a 7-point Likert-type and has a total of 40 items (1=Definitely disagree, 7=Completely agree). Cronbach's alpha coefficient for the scale is reported as 0.80-0.94.
Continued Intention to Use Scale | 6th month
  This measurement tool was developed to assess how eager individuals are to use the app. Comprises a total of 6 items and is a 7-point Likert-type (1=Definitely disagree, 7=Completely agree). There are no reversely scored items on the scale. Cronbach's alpha coefficient for the scale is reported as 0.90.
Brand Loyalty Scale | 6th month
  This scale was developed to determine the extent of individuals' loyalty to the mobile app. It comprises a total of 5 items and is a 7-point Likert-type (1=Definitely disagree, 7=Completely agree). There are no reversely scored items on the scale. Cronbach's alpha coefficient for the scale is reported as 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Topuz, PhD, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, City Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2023
Access Criteria: When this study protocol is published as an article, the link will be shared. Statistical Analysis Plan will be included in the article. The Informed Consent Form will be stored by the primary investigator. It can be requested from the researcher.

REFERENCES:
- [Background] Etbaş Demirağ H. Diabetes Risk Assessment in First Degree Relatives of Patients with Type-2 Diabetes Mellitus. T.C Adnan Menderes University Instıtute of Health Sciences, Master Thesis, 2016, Aydın, Turkey (Supervision: Prof. Dr. S Boyraz, Doç. Dr. E Ünsal Avdal).
- [Background] Turkish Society of Endocrinology and Metabolism (TEMD). Diagnosis, Treatment and Follow-up Guide for Diabetes Mellitus Complications. 14th Edition. Ankara: Bayt Publication; 2020. ISBN 978-605-4011-40-7.
- [Background] Lindstrom J, Louheranta A, Mannelin M, Rastas M, Salminen V, Eriksson J, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. The Finnish Diabetes Prevention Study (DPS): Lifestyle intervention and 3-year results on diet and physical activity. Diabetes Care. 2003 Dec;26(12):3230-6. doi: 10.2337/diacare.26.12.3230. PMID 14633807
- [Background] Martinez-Gonzalez MA, de la Fuente-Arrillaga C, Nunez-Cordoba JM, Basterra-Gortari FJ, Beunza JJ, Vazquez Z, Benito S, Tortosa A, Bes-Rastrollo M. Adherence to Mediterranean diet and risk of developing diabetes: prospective cohort study. BMJ. 2008 Jun 14;336(7657):1348-51. doi: 10.1136/bmj.39561.501007.BE. Epub 2008 May 29. PMID 18511765
- [Background] Özkan Pehlivanoğlu EF, Balcıoğlu H, Ünlüoğlu İ. The validity and reliability of the adaptation of the Mediterranean Diet Adherence Scale into Turkish. Osmangazi Medical Journal. 2020;42(2): 160-164.
- [Background] Block G, Azar KM, Romanelli RJ, Block TJ, Hopkins D, Carpenter HA, Dolginsky MS, Hudes ML, Palaniappan LP, Block CH. Diabetes Prevention and Weight Loss with a Fully Automated Behavioral Intervention by Email, Web, and Mobile Phone: A Randomized Controlled Trial Among Persons with Prediabetes. J Med Internet Res. 2015 Oct 23;17(10):e240. doi: 10.2196/jmir.4897. PMID 26499966
- [Background] McLeod M, Stanley J, Signal V, Stairmand J, Thompson D, Henderson K, Davies C, Krebs J, Dowell A, Grainger R, Sarfati D. Impact of a comprehensive digital health programme on HbA1c and weight after 12 months for people with diabetes and prediabetes: a randomised controlled trial. Diabetologia. 2020 Dec;63(12):2559-2570. doi: 10.1007/s00125-020-05261-x. Epub 2020 Sep 4. PMID 32886192
- [Background] Toro-Ramos T, Michaelides A, Anton M, Karim Z, Kang-Oh L, Argyrou C, Loukaidou E, Charitou MM, Sze W, Miller JD. Mobile Delivery of the Diabetes Prevention Program in People With Prediabetes: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 8;8(7):e17842. doi: 10.2196/17842. PMID 32459631
- [Background] Turkish Society of Endocrinology and Metabolism. (2018). Diagnosis, Treatment and Follow-up Guidelines for Diabetes Mellitus Complications, 2018.
- [Background] Roche Diagnostics Türkiye. Accu-Chek Performa Nano. Available from: www.rochediagnotics.com.tr.
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S14-S31. doi: 10.2337/dc20-S002. PMID 31862745
- [Background] Turkish Society of Endocrinology and Metabolism. Obesity Diagnosis and Treatment Guide. Ankara: Miki; 2019. ISBN: 978-605-4011-31-5.
- [Background] Hoehle H, Aljafari R, Venkatesh V. Leveraging Microsoft׳ s mobile usability guidelines: Conceptualizing and developing scales for mobile application usability. Int J Hum Comput Stud. 2016;89: 35-53.
- [Background] Güler Ç. A structural equation model to examine mobile application usability and use. International Journal of Informatics Technologies, 2019;12(3): 169-181.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT05592288/Prot_SAP_000.pdf